CLINICAL TRIAL: NCT04670497
Title: Perioperative Analgesia for Total Hip Arthroplasty: Lumbar Plexus Block Using Shamrock Technique Versus Fascia Iliaca Block
Brief Title: Perioperative Analgesia for Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Ahmed hashem, assistant lecturer at menoufia university hospital, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANET 8/2018
Record Dates: First submitted 2020-11-25; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2018-07

CONDITIONS: Regional Anesthesia
MeSH Terms: interventions — Bupivacaine; Epinephrine

STUDY DESIGN:
Intervention Model Description: This study is comparing the effect of Lumbar plexus block and fascia iliaca block with general anesthesia to provide perioperative pain control and compare their effects on hemodynamics.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: sealed opaque envelop
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasound guided lumbar plexus block (Active Comparator): patients were recieved lumbar plexus block ultrasound guided by shamrock technique using 0.5% bupavacaine in a dose 0.3ml/kg
  Interventions: Procedure: bupivacaine 0.5% with 1:200000 adrenaline
- ultrasound guided Fascia iliaca block (Active Comparator): patients were received fascia iliaca block ultrasound guided using 0.5% bupoavacaine in a dose 0.3ml\kg
  Interventions: Procedure: bupivacaine 0.5% with 1:200000 adrenaline

INTERVENTIONS:
Procedure: bupivacaine 0.5% with 1:200000 adrenaline — regional anesthesia to block lumbar plexus for analgesia of lower limb

SUMMARY:
This study is comparing the effect of lumbar plexus block and fascia iliaca block with general anesthesia to provide perioperative pain control and compare their effects on hemodynamics

DETAILED DESCRIPTION:
Different groups receive different interventions at same time during study. patients were randomly allocated in two groups :

Group A: lumbar plexus block using shamrock technique by 0.3 ml/kg of 0.5% bupivacaine with 1:200000 adrenaline.

Group B: Fascia iliaca block by 0.3 ml/kg of 0.5% bupivacaine with 1:200000 adrenaline.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II and scheduled for elective total hip arthroplasty

Exclusion Criteria:

* Patients who refuse to participate.
* Local infection.
* Patients with coagulation defects

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Assessment of postoperative analgesia | 24 hours
  each patient was assessed by visual analogue scale which consists of a 10 cm line with one end labelled "no pain" and the other end labelled "worst pain imaginable". The patient marks the line at the point that best describes the pain intensity

SECONDARY OUTCOMES:
Compare effects of both groups on mean arterial blood pressure | intraoperative and 24 hours
  monitoring of blood pressure using non invasive blood pressure measurement in millimeter mercury

OTHER OUTCOMES:
compare their effects on heart rate (beat\minute) | intraoperative and 24 hours
  monitoring of heart rate using pulse oximetry in beat\minute
Complication rate for procedures in the form of local anesthetic toxicity | Intraoperative monitoring
  observation of occurrence of local anesthetic toxicity as hypotension, seizures, bradycardia

CONTACTS AND LOCATIONS:
Overall Officials: ahmed abd elraof, professor, Study Chair — faculty of medicine, anesthesia department; Ezz elden saleh, professor, Study Chair — faculty of medicine, anesthesia department; sadek abdelmasih, lecturer, Study Director — faculty of medicine, anesthesia department
Locations (1):
- Ahmed hashem, Cairo, Assistant Lecturer, Egypt

IPD SHARING:
Plan to Share IPD: No